CLINICAL TRIAL: NCT05054101
Title: Life With Covid Since 2020: a Randomized Control Trial of a Real-time Data Collection Smartphone-based App Assessing and Treating the Covid-19 Psychological Impacts
Acronym: VieCovid2020
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unresolved issues between research partners (research has not started)
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: APHP200426; 2021-A02141-40 (Other: IDRCB)
Record Dates: First submitted 2021-09-22; First posted 2021-09-23 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VieCovid2020 smartphone application (Experimental): The VieCovid2020 smartphone application in add-on to usual psychiatric intervention
  Interventions: Other: Real-time assessment using the VieCovid2020 smartphone application
- Usual psychiatric intervention (Placebo Comparator): Usual psychiatric intervention alone
  Interventions: Other: Real-time assessment using the VieCovid2020 smartphone application

INTERVENTIONS:
Other: Real-time assessment using the VieCovid2020 smartphone application — a real-time assessment using the VieCovid2020 smartphone application during the first 3 months in add-on to usual psychiatric intervention

SUMMARY:
The COVID-19 pandemic and more specifically the confinement is an unpleasant experience for those who undergo it. Separation from loved ones, the loss of freedom, uncertainty over disease status, and boredom can, on occasion, create dramatic effects.

In fact, the pandemic and its consequences are inducing a considerable degree of fear, worry and concern in the population at large and among certain groups in particular, such as older adults, care providers and people with underlying health conditions.

If we refer back to former pandemics (SARS-CoV-1, MERS, Ebola), suicide, post-traumatic stress disorder (PTSD) and adjustment disorders have been reported, anger generated, and lawsuits brought.

The current COVID-19 pandemic is an epidemiological and psychological crisis. The enormity of living in isolation, changes in our daily lives, job loss, financial hardship and grief over the death of loved ones has the potential to affect the mental health and well-being of many.

Given the developing situation with Covid-19, policy makers urgently need evidence synthesis to produce guidance for the public and patients suffering from mental disorders such as PTSD and adjustment disorders. Therefore, it seems crucial to assess and manage the signs of anxiety, panic attacks, depression and suicide easily and at the national scale using fast, efficient and cutting-edge techniques.

Objectives :

To assess the superiority of the VieCovid2020 smartphone app, in add-on to usual care in patients suffering from PTSD or adjustment disorders within the context of COVID-19, on the rate of responders at 6 months using the PCL-5 (PTSD Checklist for DSM-5)

The VieCovid2020 smartphone application provides lifestyle and educational advices, as well as, a real-time data collection targeted the emotional state of the user.

It will be used during 3 months in add-on to usual psychiatric intervention and psychiatric evaluations.

DETAILED DESCRIPTION:
Design of the study :

Multicentric randomized controlled superiority trial with 2 parallel arms. The randomization will be a various-sized block randomization, stratified by centre and by co-treatment (=usual psychiatric intervention) prescribed at baseline before randomisation: selective serotonin reuptake inhibitors (SSRI) alone or SSRI in combination to eye movement desensitization and reprocessing (EMDR), cognitive behavioural therapy (CBT) or reconsolidation blockade.

Objectives :

To assess the superiority of the VieCovid2020 smartphone app, in add-on to usual care in patients suffering from PTSD or adjustment disorders within the context of COVID-19, on the rate of responders at 6 months using the PCL-5 (PTSD Checklist for DSM-5)

Every patient will be randomized between:

* usual psychiatric intervention alone and psychiatric evaluations at 5 following time points (day 1, 1 month, 3 months, 6 months and 12 months) (control arm) or
* a real-time assessment using the VieCovid2020 smartphone application during the first 3 months in add-on to usual psychiatric intervention and psychiatric evaluations at 5 following time points (day 1; 1 month; 3 months, 6 months and 12 months) (intervention arm)

Use of the VieCovid2020 smartphone application and psychiatric evaluations at 5 following time points are added by the research.

Population :

Volunteers suffering from PTSD or adjustment disorders will be included within the study.

Application :

The VieCovid2020 smartphone application provides lifestyle and educational advices, as well as, a real-time data collection targeted the emotional state of the user.

It will be used during 3 months in add-on to usual psychiatric intervention and psychiatric evaluations.

Expected benefits :

A potential reduction of acute and chronic stress is expected among users of the application in particular with the set of lifestyle and educational advices proposed every week.

In the COVID-19 pandemic context, the expected benefits for society is to contribute to reduce the number of patients suffering from PTSD or adjustment disorders.

850 patients are expected and 18 sites in France.

ELIGIBILITY:
Inclusion criteria :

* PTSD or adjustment disorders criteria according to DSM-5 and MINI criteria within the context of COVID-19 trauma exposure and economic consequences;
* patients with a PCL-5 score higher than 33;
* patient treated or who will be treated by the following treatments: SSRIs alone or SSRIs in combination to CBTs, EMDR or reconsolidation blockade
* able to download and use an app, with a correct internet connection (owner of a smartphone)
* Affiliation to a French social security system (recipient or assign) excluding AME
* written consent to participate in the study;

Exclusion criteria :

* age lower than 18, without any upper age limit;
* suicidal risk using MINI;
* non-French speaker;
* guardianship curatorship and person deprived of their liberty by judicial decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Superiority of the VieCovid2020 smartphone app | 6 MONTHS
  To assess the superiority of the VieCovid2020 smartphone app, in add-on to usual care in patients suffering from adjustments disorders or PTSD within the context of COVID-19, on the rate of responders at 6 months on the PCL-5.

SECONDARY OUTCOMES:
User adherence of the VieCovid app | 3 months
  To assess the user adherence of the VieCovid2020 smartphone application at 3 months
Impact of co-treatments | 3 months
  To assess the impact of co-treatments on superiority of the VieCovid2020 smartphone app, in add-on to usual care in patients suffering from adjustments disorders or PTSD within the context of COVID-19, on the rate of responders on the PCL-5 at 3, 6 and 12 months .
Economic Impact | 6 months
  To assess the economic impact of using the VieCovid2020app